CLINICAL TRIAL: NCT05628493
Title: Gut Microbiota Analysis With Next-generation 16S rRNA Gene Sequencing in IAI Patients With Sepsis-associated Liver Dysfunction
Brief Title: Gut Microbiota Analysis in IAI Patients With Sepsis-associated Liver Dysfunction
Acronym: 2022-11-09
Status: Completed | Type: Observational
Sponsor: Chinese Medical Association (Network)
Responsible Party: Sponsor
Other Study IDs: 2022-11-09
Record Dates: First submitted 2022-11-09; First posted 2022-11-28 (Actual); Last update posted 2022-11-28 (Actual); Status verified 2022-03

CONDITIONS: Gut Microbiota; Intra-abdominal Infections; Acute Gastrointestinal Injury; Sepsis-associated Liver Dysfunction
MeSH Terms: conditions — Intraabdominal Infections

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Patient Registry: Yes
Target Follow-Up Duration: 28 Days
Biospecimen Retention: Samples With DNA — fecal samples were collected per patient on days 1,3 and 7 after ICU admission. All fecal samples were collected in sterile tubes and then stored at -80°C refrigerator.
  The gut microbiota analysis was performed by LC-Bio Technology Co., Ltd. (Hangzhou, China)
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- The non-SALD group: The patient did not meet the SALD diagnosis during the study observation period. SALD was diagnosed when the level of serum alanine aminotransferase (ALT) or aspartate aminotransferase (AST) ≥ 1000IU/L, or total bilirubin (TBIL) level >3mg/dL during hospitalization.
  Interventions: Behavioral: Gut microbiota Analysis
- The SALD group: The patient's maximum values of ALT, AST, or TBIL during hospitalization reached any of the SALD criteria.
  Interventions: Behavioral: Gut microbiota Analysis

INTERVENTIONS:
Behavioral: Gut microbiota Analysis — fecal samples were collected per patient on days 1,3 and 7 after ICU admission. All eligible patients were given antibiotics therapy, actively control infection source by puncture drainage or surgery if necessary, as well as other supportive therapy to maintain organ function.

SUMMARY:
With the rapid development of intensive care medicine, the mortality of patients with sepsis has decreased over the past decade, but it is still the leading cause of death in intensive care unit (ICU). As an important immune and metabolic organ, the liver plays a crucial role in host defense against invading pathogens and endotoxins, as well as maintenance of metabolic and immunological homeostasis. Some studies indicate that sepsis-associated liver dysfunction (SALD) has a substantial impact on the severity and prognosis of sepsis.

Intra-abdominal infections (IAI) are the second leading source of infection for sepsis after pneumonia in ICU, and are often related to high morbidity and mortality rates. Studies had found that the incidence of SALD in IAI patients was considerably higher than that of general population with sepsis. Moreover, the incidence of acute gastrointestinal injury (AGI) in IAI patients was also much higher than that in sepsis patients with other site infections, as well as the degree of AGI was more serious according to guidelines proposed by the European Society of Intensive Care Medicine (ESICM) in 2012. IAI can directly cause AGI, and a subset of patients usually progress to increased intra-abdominal pressure, which further aggravates AGI.

The pathogenesis of SALD remains unclear so far, and its mechanism is complicated and elusive. Nevertheless, the unique anatomical structure of the liver make it has close association with the gut, growing evidence indicates that the gut microbiota and related metabolites are related to several liver disease. In case of sepsis, gut microbiota disorder and low microbial diversity can cause severe liver injury. An important mechanism for this phenotype is the gut-liver axis, which refers to gut microbial metabolites and nutrients are transported to the liver through the portal vein and hepatic artery to maintain the healthy metabolism of liver.

Therefore, we initially conducted a retrospective study to investigate the relationship between the occurrence of AGI and SALD among IAI patients. Subsequently, a prospective study was performed to analyze and compare the diversity and composition of gut microbiota in IAI patients with or without SALD, respectively, and the dynamic changes in the gut microbiota during the first week after ICU admission were also investigated.

DETAILED DESCRIPTION:
A retrospective cohort study was conducted involving sepsis patients with IAI treated in ICU department of Nanjing Drum Tower Hospital between April 2020 to April 2020. Adult patients (≥18 years) with IAI who met the criteria for sepsis 3.0 were included. The exclusion criteria included: discharged or died within 48 hours after ICU admission; known serious chronic liver disease, such as decompensated cirrhosis and end-stage liver cancer; hospitalization due to primary hepatobiliary disease, such as trauma, hepatitis, cholelithiasis, etc; other causes of liver injury include: drugs, poisons, etc; and pregnancy.The following data were collected within 24 hours after ICU admission: demographic Information: age, sex and comorbidity; the score of disease severity: Acute Physiology and Chronic Health Evaluation (APACHE) II score; Sequential Organ Failure Assessment (SOFA) score; the primary site of abdominal infection: upper or lower gastrointestinal tract, pancreas and others; laboratory indicators: white blood cells (WBC), percentage of neutrophils (N%), C-reactive protein (CRP), procalcitonin (PCT), human leukocyte antigen (HLA)-DR. Date during hospitalization were also collected: complications: respiratory failure, septic shock, acute kidney injury (AKI) and AGI; pathogenic bacteria of ascites culture; bacteremia or not; total parenteral nutrition (TPN) was given or not. Prognostic indicators included ICU length of stay (LOS), hospital LOS, ICU mortality, in-hospital mortality, and 28-day mortality were also recorded.SALD was diagnosed when the level of serum alanine aminotransferase (ALT) or aspartate aminotransferase (AST) ≥ 1000IU/L, or total bilirubin (TBIL) level >3mg/dL during hospitalization. IAI was diagnosed according to the 2005 International Sepsis Forum Consensus Conference. Briefly, the patient present with abdominal symptoms and signs, such as fever (≥38℃), tenderness, rebound pain, etc; elevated inflammatory indicators in peripheral blood and positive culture of intra-abdominal specimens. Sepsis 3.0 and septic shock were diagnosed according to Third International Consensus Definition for Sepsis and Septic Shock in 2016. AKI was diagnosed according to the Kidney Disease Improving Global Outcomes (KDIGO) clinical practice guidelines. AGI diagnosis and grading are based on the ESICM recommendations in 2012.To further clarify the relationship between gut microbiota and SALD, we conducted a prospective observational study between April 2020 to April 2020 in our center. Eligible patients must fulfill the same criteria as above. Other exclusion criteria also include: with expected ICU LOS < 1 week; had participated in any other clinical trial; underwent enterostomy surgery; had chronic inflammatory bowel disease. All eligible patients were given antibiotics therapy, actively control infection source by puncture drainage or surgery if necessary, as well as other supportive therapy to maintain organ function. Moreover, fecal samples were collected per patient on days 1,3 and 7 after ICU admission. Other data collection and the definition of related diseases are the same as the above.

ELIGIBILITY:
Inclusion Criteria:

* Adult patients (≥18 years)
* Diagnosed as Intra-abdominal infections (IAH)
* Diagnosed as sepsis 3.0

Exclusion Criteria:

* Discharged or died within 48 hours afterenrollment
* Known serious chronic liver disease, such as decompensated cirrhosis and end-stage liver cancer
* Hospitalization due to primary hepatobiliary disease, such as trauma, hepatitis, cholelithiasis, etc;
* Other causes of liver injury include: drugs, poisons, etc
* Pregnancy.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All patients diagnosed with intra-abdominal infection (IAI). IAI was diagnosed according to the 2005 International Sepsis Forum Consensus Conference. Briefly, the patient present with abdominal symptoms and signs, such as fever (≥38℃), tenderness, rebound pain, etc; elevated inflammatory indicators in peripheral blood and positive culture of intra-abdominal specimens.
Sampling Method: Non-Probability Sample
Enrollment: 20 (Actual)
Dates: Start 2022-01-03 (Actual); Primary Completion 2022-09-09 (Actual); Study Completion 2022-09-14 (Actual)

PRIMARY OUTCOMES:
mortality | Day28 after enrollment
  28day-mortality

SECONDARY OUTCOMES:
Gastrointestinal function | through study completion, an average of 7 days
  acute gastrointestinal injury (AGI)
Gut microbiota | days 1,3 and 7 after enrollment
  analysis of gut microbiota by 16S rRNA sequencing

CONTACTS AND LOCATIONS:
Overall Officials: Wenkui Yu, Ph.D., Study Chair — Study concept and study design
Locations (1):
- Nanjing Drum Tower Hospital, Nanjing, Jiangsu, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Guo K, Ren J, Wang G, Gu G, Li G, Wu X, Chen J, Ren H, Hong Z, Wu L, Chen G, Youming D, Li J. Early Liver Dysfunction in Patients With Intra-Abdominal Infections. Medicine (Baltimore). 2015 Oct;94(42):e1782. doi: 10.1097/MD.0000000000001782. PMID 26496306
- [Result] Yang XJ, Liu D, Ren HY, Zhang XY, Zhang J, Yang XJ. Effects of sepsis and its treatment measures on intestinal flora structure in critical care patients. World J Gastroenterol. 2021 May 21;27(19):2376-2393. doi: 10.3748/wjg.v27.i19.2376. PMID 34040329